CLINICAL TRIAL: NCT01856842
Title: Reperfusion of Pulmonary Arteriovenous Malformations After Embolotherapy. A Randomized Trial of Interlock™ Fibered IDC™ Occlusion System vs. Nester Coils
Brief Title: Reperfusion of Pulmonary Arteriovenous Malformations After Embolotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01-ANGIO-12
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Arteriovenous Malformations
Keywords: Pulmonary Arteriovenous Malformations; Hereditary Hemorrhagic Telangiectasia (HHT); Embolization; reperfusion rates
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interlock fibered IDC Occlusion System (Active Comparator): Pulmonary angiography and embolotherapy technique using Interlock (TM) fibered IDC Occlusion System(TM)
  Interventions: Procedure: Angiography and embolotherapy
- Nestor Coil (Active Comparator): Pulmonary angiography and embolotherapy technique using Nestor coils
  Interventions: Procedure: Angiography and embolotherapy

INTERVENTIONS:
Procedure: Angiography and embolotherapy

SUMMARY:
AVMs are abnormal collections of blood vessels which can occur in any part of the body including the lungs. These blood vessels are weakened and can rupture anytime causing bleeding which can be massive, leading to life-threatening conditions.

Pulmonary AVMs occur in about 40% of patients with HHT. Each patient may have an average of 5 AVMs .Rupture of the AVM can lead to massive bleeding in the lung, stroke and infection of the brain. In order to prevent these complications, patients with HHT are routinely examined for pulmonary AVMs and treatment with embolization is recommended.

AVMs have a main blood vessel or artery supplying blood to the collection of blood vessels. The way to treat AVMs is cut off their blood supply through a process called embolization.

Embolization is a standard medical procedure which is done to stop or prevent hemorrhage (bleeding) from an AVM. It involves blocking the artery that supplies blood to the AVM by inserting a foreign body, into the blood vessel supplying blood to the AVM.

Standard devices used for embolization include coils (made of stainless steel or platinum). These devices usually have a good success rate for blocking the artery that supplies blood to the AVM. However, a few AVMs that are embolized by standard devices may reopen over time. This is called reperfusion and will require repeat embolization procedures.

For embolization of pulmonary AVMs at St. Michael's Hospital, the Nester coil is used. In this study, we would like to compare the Nester coil with a new coil device called the Interlock Fibered IDC Occlusion System. Both coils are approved for use in Canada, however the cost of the IDC coil limits its use at this hospital.

Compared to the Nester coil, the IDC coils are made so that they can be removed or repositioned if they are not placed correctly. The coil also allows tighter packing which helps prevent reperfusion.

This study will compare the success rate of embolization between the Interlock™ Fibered IDC™ Occlusion System (IDC coil) and the Nester coil.

DETAILED DESCRIPTION:
Introduction Pulmonary arteriovenous malformations (AVMs) can lead to life-threatening complications. These complications can be prevented with pre-symptomatic embolization. The Interlock™ Fibered IDC™ Occlusion System coil (IDC) is a new device which might be more effective for embolizing pulmonary AVMs. This study will investigate the efficacy of the Interlock™ Fibered IDC™ Occlusion System and compare rates of reperfusion using Nestor coils (standard coils used at participating centre) versus Interlock™ Fibered IDC™ Occlusion, randomizing by AVM.

Rationale Reperfused AVMs put the patient at risk of pulmonary AVM complications. As such, these AVMs require repeat embolotherapy and therefore patients are subjected to further radiation, contrast and hospitalization. A number of devices have been studied and are currently being used for embolization of pulmonary AVMs including coils (stainless steel, platinum) and plugs (Amplatzer plugs). The immediate technical success rate is nearly 100%, but long-term reperfusion occurrence is approximately 15% of treated AVMs and up to 30% of patients. The IDC coil characteristics may lead to reduced reperfusion rates. No studies of IDC coils have been reported to date in the management of pulmonary AVMs. Safety of IDC coils has been demonstrated in other organs. Embolization procedure with IDC coils is similar to embolization with other devices, in terms of fluoroscopy time use and contrast load, as are procedural complication rates.

Background Pulmonary AVMs are present in approximately 40% of patients with hereditary hemorrhagic telangiectasia (HHT), with a mean of five pulmonary AVMs per patient. Pulmonary AVMs can lead to life-threatening and debilitating complications, such as massive haemoptysis, spontaneous haemothorax, stroke and cerebral abscess. Fortunately, these complications are preventable, through screening of HHT patients and preventative treatment of pulmonary AVMs, as summarized in a recent decision analysis. The International HHT Guidelines recommends routine screening of all HHT patients for pulmonary AVMs, with preventative transcatheter embolotherapy of all significant pulmonary AVMs.

Most published data have reported outcomes with stainless steel or platinum coils, and fewer with detachable balloons or Amplatzer plugs. Even with good success rates, reperfusion has generally been reported in the range of 15% of embolized AVMs with routine embolization using stainless steel or platinum coils. To date, comparative studies between stainless steel and platinum coils have not shown significant differences in outcomes.

PLAN OF INVESTIGATION Study Hypothesis The device of interest has local characteristics including better positioning and controlled release, together with tighter packing, which may lead to superior outcomes and reduce costs as well as radiation time. Therefore it is hypothesized that the IDC coil will be associated with less reperfusion than standard Nestor coils, and will present a therapeutic advantage over Nestor coils.

Objectives Primary Objective Reperfusion for each AVM will be assessed at 1-year follow-up post-embolization. If there is insufficient involution (<70% by volume) of the lesion, then the AVM will be considered to be reperfused and care will be according to best clinical practice. Follow up imaging will be as per usual practice/guidelines. If the participant develops complications suspected to be due to pulmonary AVMs during the first year follow-up period, then reassessment will be arranged according to current clinical practice protocols. If there is evidence at early follow-up of ongoing AVM perfusion or of lack of aneurismal involution, the AVM will be considered to be "reperfused".

Secondary Objective Reported secondary outcomes include fluoroscopy time, contrast volume required, procedural time and complication rates.

STUDY DESIGN Study Population All adult patients who attend the Hereditary Hemorrhagic Telangiectasia (HHT) clinic, require embolization procedures for their pulmonary AVMs, who meet the inclusion and exclusion criteria will be considered eligible for this study. The Toronto HHT Centre has a large well-characterized HHT population (approximately 1000 patients), the largest such population in Canada, allowing for feasible recruitment. It is estimated that approximately 30 new patients undergo embolization per year, comprising approximately 150 AVMs.

Enrollment Potential study participants will be identified from the Toronto HHT Centre Database, an IRB approved comprehensive database capturing clinical information of patients who have expressed an interest to participate in HHT related research studies and/or from the HHT Clinic. Potential participants will be pre- screened for eligibility and upon determination be approached for study participation. The study will initially be presented to the eligible patient by the treating physician or a member of the HHT clinic team, who will then introduce study personnel to the patient in order to give any additional information including obtaining informed consent.

Randomization

Each participant will receive a unique randomization list. The Investigators will first determine the number of pulmonary AVMs for which embolotherapy is required per participant. Each treatable AVM will be referenced anatomically and assigned a number starting from one and continuing up in sequential order. The Study Coordinator will then match this list to a pre determined randomization list. Each AVM will be randomized into one of the two following treatment allocations:

1. AVM Allocation I: Standard embolization procedure with Nestor Coil
2. AVM Allocation II: Standard embolization procedure with The Interlock™ Fibered IDC™ Occlusion System coil Unused randomizations will be discarded and will not be carried over to the subsequent enrolled participant. The Investigators will not have access to the randomization lists but will be informed by the Study Coordinator as to which AVM will acquire which allocated treatment device.

Blinding

Blinding of the Principal Investigator is not possible since the Primary Investigator is also the treating Interventional Radiologist responsible for the embolotherapy procedure. Participants will be blinded to the type of coil they receive (Group Allocation) for each particular treatable aneurysm. Outcome ascertainment bias will be minimized by the following:

1. Coil allocation will be performed by the Study Coordinator during randomization
2. Final analysis results are non-subjective and obtained from concrete values acquired from imaging data such as reperfusion rate per coiled aneurysm

STUDY VISITS Visit I - Screening and Baseline The study will be explained in detail to the eligible participant. They will be given as much time as needed to review the informed consent form (ICF) and ask any questions they may have regarding the study. It will be ensured that all questions regarding the study are answered to satisfaction of the eligible participants.

Once satisfied and prior to commencement of any study related procedures, the participant will be asked to sign the Research Ethics Board-approved written consent form for this study. A copy of the informed consent form will be provided to the patient to take and look over at their leisure.

After informed consent is obtained, the Study Coordinator will screen patients for study eligibility using the inclusion/exclusion criteria defined in this protocol and will document them on a screening log. Reasons for non-participation will be identified based on inclusion and exclusion criteria.

Visit II - Procedure Pulmonary angiography and embolotherapy will be performed using standard clinical technique. Using standard aseptic technique the right common femoral vein is punctured under direct sonographic guidance. A 7 French sheath is placed and connected to a continuous saline irrigation. The right heart and then pulmonary arteries cannulated using a 7 French Van Aman catheter. Pulmonary artery pressures are obtained; followed by pulmonary angiography, either unilateral or bilateral depending on the site of the PAVMs. Once confirmed the feeding arteries are cannulated using the Lumax catheter. After confirming position the coils are deployed until complete occlusion of the feeding artery is achieved. Similar procedure repeated for the other PAVMs. The catheter and sheath are then removed and haemostasis is obtained. The participant is sent to the ward for monitoring.

Visit III - Post Procedure Post procedure, the participant will follow standard clinical practice recommendations. The participant will be admitted overnight and will undergo a routine chest X-Ray 1-day post embolization, before discharge from the hospital. The participant will be assessed for the presence of post-procedure complications.

Visit IV - Month 1-3 Follow-Up As per standard clinical practice, the participant will be required to visit Dr. Faughnan at the HHT Clinic 1-3 months post-procedure. This visit will also include a single view chest X-Ray and standard oxygen shunt test. If there is any suspicion of reopening of the embolized artery, it will be managed as per usual clinical practice.

Visit V - Month 10-14 Follow-Up As per usual clinical practice, the participant will be re-assessed at 10-14 months post-procedure with an unenhanced low-dose CT scan of the chest. If there is any suspicion of reopening of the embolized artery, this will be managed as per usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for inclusion in the study if all the following criteria are met:

1. Documented presence of new (untreated) pulmonary AVMs requiring embolization
2. Definite clinical diagnosis of HHT or genetic diagnosis of HHT
3. Age ≥18 years
4. Able to provide informed consent

Exclusion Criteria:

Patients will be excluded from the study if, in the opinion or knowledge of the Principal Investigator any of the following criterion is present:

1. Participants with multiple AVMs within close proximity where identification of the aneurysm seen on CT cannot be precisely isolated for randomization purposes.
2. Contra-indications to embolotherapy

   1. Severe chronic renal failure, without availability of dialysis
   2. Severe pulmonary hypertension (PA systolic estimated at >60mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Difference in reperfusion rate | 10-14 months post embolization
  The primary end-point for this study is the difference in reperfusion rate between the two treatment groups from procedure day to the final follow-up at 10-14 month post embolization, measured by the unenhanced CT Chest.

SECONDARY OUTCOMES:
Fluoroscopy/radiation time | during procedure
  Fluoroscopy/radiation time
Contrast volume required | during embolization
  Contrast volume required
Procedural time | during embolization
  Procedural time
Complication rates | during embolization
  Complication rates
Cost analysis | during 10-14 months post procedure that is to final visit
  Cost analysis

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Prabhudesai, MD, Principal Investigator — Unity Health Toronto; Marie Faughnan, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kennedy SA, Faughnan ME, Vozoris NT, Prabhudesai V. Reperfusion of Pulmonary Arteriovenous Malformations Following Embolotherapy: A Randomized Controlled Trial of Detachable Versus Pushable Coils. Cardiovasc Intervent Radiol. 2020 Jun;43(6):904-909. doi: 10.1007/s00270-020-02422-8. Epub 2020 Feb 4. PMID 32020296